CLINICAL TRIAL: NCT03849846
Title: Recruiting Participants With Low Socioeconomic Status in the NutriQuébec Study: Using Focus Groups to Explore Their Beliefs, Preferences and Concerns
Brief Title: Using Focus Groups to Explore Perceptions of Adults With Low Socioeconomic Status Regarding the NutriQuébec Study
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-042 A-1/18-05-2018
Record Dates: First submitted 2019-01-10; First posted 2019-02-21 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Focus Groups
Keywords: Low socioeconomic status population; Web-based prospective cohort study; Focus groups; Recruitment; Behavioural beliefs; Normative beliefs; Control beliefs; Security of data; Use of data; Share of data
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with low socio-economic status: Four focus groups will be conducted with adults with low socioeconomic status recruited through community centres in the Québec City area.
  Interventions: Other: Focus groups

INTERVENTIONS:
Other: Focus groups — Participants will also complete a sociodemographic questionnaire. The moderator will conduct the discussion using a semi-structured interview guide, based on the construct of the Theory of Planned Behaviour. The interview guide has been developed to identify the beliefs that determine the participants' attitudes (advantages/disadvantages), subjective norms (approval/disapproval of important others) and perceived behavioural control (facilitators/barriers) related to a hypothetical participation in the NutriQuébec study. The participants will also be questioned about their preferences regarding the recruitment as well as their concerns about the security, use and share of data.

SUMMARY:
NutriQuébec is a web-based prospective cohort study aiming to monitor and analyse the evolution of Québec population eating habits through annual questionnaires. The recruitment and retention of participants with low socioeconomic status (SES), known to be more hard to reach and recruit into health studies, will be major challenges in obtaining a representative sample of the Québec population.

The purpose of this study is to identify the behavioural, normative and control beliefs of individuals from low SES regarding a hypothetical participation in the NutriQuébec study. Their preferences regarding recruitment methods as well as their concerns about the security, use and share of data will also be identified.

Four moderator facilitated focus groups will be conducted in community centres (n=28 participants). The focus groups will be recorded, transcribed and coded by two coders using NVivo.

DETAILED DESCRIPTION:
Four focus groups will be conducted in three community centers (n=6 to 8 participants/group; n=28 participants). First, all participants will read and sign the consent form. They will also complete a sociodemographic questionnaire. Then, the moderator will conduct the discussion using a semi-structured interview guide, based on the construct of the Theory of Planned Behaviour. The interview guide has been developed to identify the beliefs that determine the participants' attitudes (advantages/disadvantages), subjective norms (approval/disapproval of important others) and perceived behavioral control (facilitators/barriers) related to a hypothetical participation in the NutriQuébec study. The participants will also be questioned about their preferences regarding the recruitment as well as their concerns about the security, use and share of data. The focus groups will be recorded and transcribed. Two coders will perform the codification independently using NVivo 10.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age and older)
* Living in the Québec City Metropolitan Area
* Attending one of the three community centers where the focus groups will be conducted
* Be able to answer questionnaires in French

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with low socioeconomic status
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
The perceived advantages related to a hypothetical participation in the NutriQuébec study is based on the Theory of Planned Behaviour (behavioural beliefs) and will be identified from focus groups. | Baseline
  The perceived advantages related to a hypothetical participation in the NutriQuébec study is based on the Theory of Planned Behaviour (behavioural beliefs) and will be identified from focus groups. The question asked to participants will be: In your opinion, what would be the advantages of participating in the NutriQuébec study?
The perceived disadvantages related to a hypothetical participation in the NutriQuébec study is based on the Theory of Planned Behaviour (behavioural beliefs) and will be identified from focus groups. | Baseline
  The perceived disadvantages related to a hypothetical participation in the NutriQuébec study is based on the Theory of Planned Behaviour (behavioural beliefs) and will be identified from focus groups. The question asked to participants will be: In your opinion, what would be the disadvantages of participating in the NutriQuébec study?
The persons most likely to approve the participant hypothetical participation in the NutriQuébec study is based on the Theory of Planned Behaviour (normative beliefs) and will be identified from focus groups. | Baseline
  The persons most likely to approve the participant hypothetical participation in the NutriQuébec study is based on the Theory of Planned Behaviour (normative beliefs) and will be identified from focus groups.
  The question asked to participants will be: Among the people (groups or individuals) important to you, which ones would agree that you should participate in the NutriQuébec study? For what reasons?
The persons most likely to disapprove the participant hypothetical participation in the NutriQuébec study is based on the Theory of Planned Behaviour (normative beliefs) and will be identified from focus groups. | Baseline
  The persons most likely to disapprove the participant hypothetical participation in the NutriQuébec study is based on the Theory of Planned Behaviour (normative beliefs) and will be identified from focus groups. The question asked to participants will be: Among the people (groups or individuals) important to you, which ones would not agree with the fact that you are participating in the NutriQuébec study? For what reasons?
The facilitators related to a hypothetical participation in the NutriQuébec study is based on the Theory of Planned Behaviour (control beliefs) and will be identified from focus groups. | Baseline
  The facilitators related to a hypothetical participation in the NutriQuébec study is based on the Theory of Planned Behaviour (control beliefs) and will be identified from focus groups. The question asked to participants will be: In your opinion, what would help you participate in the NutriQuébec study?
The barriers related to a hypothetical participation in the NutriQuébec study is based on the Theory of Planned Behaviour (control beliefs) and will be identified from focus groups. | Baseline
  The barriers related to a hypothetical participation in the NutriQuébec study is based on the Theory of Planned Behaviour (control beliefs) and will be identified from focus groups. The question asked to participants will be: In your opinion, what would prevent you from participating in the NutriQuébec study?

SECONDARY OUTCOMES:
The preferences about the recruitment in the NutriQuébec study will be identified from focus groups. | Baseline
  The preferences about the recruitment in the NutriQuébec study will be identified from focus groups. The question is: What ways would be effective to recruit you into the NutriQuébec study? If we advertised the NutriQuébec study, how could you hear about us?
The concerns about the security of the data in the NutriQuébec study will be identified from focus groups. | Baseline
  The concerns about the security of the data in the NutriQuébec study will be identified from focus groups. The question is: Do you have any concerns about the security of the data that will be collected using the web questionnaires?
The concerns about the use of the data in the NutriQuébec study will be identified from focus groups. | Baseline
  The concerns about the use of the data in the NutriQuébec study will be identified from focus groups. The question is: Do you have any concerns about the use and sharing of data between different researchers, knowing that they will not have access to your personal data such as your name and health insurance number?
The concerns about the share of the data in the NutriQuébec study will be identified from focus groups. | Baseline
  The concerns about the share of the data in the NutriQuébec study will be identified from focus groups. The question is: Do you have any concerns about the use and sharing of data between different researchers, knowing that they will not have access to your personal data such as your name and health insurance number?

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Canada

IPD SHARING:
Plan to Share IPD: No